CLINICAL TRIAL: NCT05097872
Title: Targeted Elimination Diet in IBS Patients Following Identification of Trigger Nutrients Using Confocal Laser Endomicroscopy
Brief Title: ConfocAl endomicroSCopy bAsed Diet Trial in IBS
Acronym: CASCADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S65495
Record Dates: First submitted 2021-10-15; First posted 2021-10-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Real diet (Active Comparator): Diet excluding the trigger nutrient identified by an acute mucosal reaction in CLE
  Interventions: Other: Diet
- Sham diet (Sham Comparator): Diet excluding a sham nutrient without acute mucosal reaction in CLE
  Interventions: Other: Diet
- Wheat exclusion diet (Active Comparator): In patients without identified trigger nutrient (i.e. no acute mucosal reaction to any nutrient), wheat will be excluded as an empirical diet in crossover fashion with soy.
  Interventions: Other: Diet
- Soy exclusion diet (Active Comparator): In patients without identified trigger nutrient (i.e. no acute mucosal reaction to any nutrient), wheat will be excluded as an empirical diet in crossover fashion with soy.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Diet excluding either trigger and sham nutrient in a blinded crossover fashion (CLE positive individuals with identified trigger) or wheat and soy in a blinded crossover fashion (CLE negative individuals without identified trigger)

SUMMARY:
After a thorough baseline evaluation, IBS patients will be exposed to nutrients while undergoing confocal laser endomicroscopy (CLE). Patients presenting an acute mucosal reaction upon nutrient exposure will be instructed to exclude their respective trigger nutrient or a nutrient without mucosal reaction (=sham diet) from their diet for 4 weeks in a randomized, blinded crossover fashion.

The aim of the trial is to assess the symptomatic response to the targeted diet and further elucidate mechanisms underlying the acute mucosal reactions observed in CLE upon nutrient exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 y/o (70 years included)
* Male or female subjects
* IBS-D and IBS-M (i.e. IBS-non-C) according to Rome IV criteria
* Moderate to severe symptom severity as defined by the Irritable bowel syndrome severity scoring system (IBS-SSS) (i.e. IBS-SSS >175 points)
* Provide written informed consent to participate in the study
* Women of child-bearing potential agree to apply a highly effective method of birth control during the entire duration of the trial. Highly effective birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.
* Subjects who are capable to understand the study and the questionnaires, and to comply with the study requirements.

Exclusion Criteria:

* - Pregnant or breastfeeding women
* History of major surgery of the gastrointestinal tract (cholecystectomy and uncomplicated appendectomy are allowed)
* Symptoms predominantly associated with functional dyspepsia or gastro-esophageal reflux disease
* Immunoglobuline E (IgE)-mediated food allergies identified by immunocap blood tests or skin prick testing
* Known underlying organic gastrointestinal disease
* Current or recent use of NSAIDs, proton-pump inhibitors, systemic histamine-receptor antagonists, mast cell stabilizers, corticosteroids, opioids (need to be stopped at least 2 weeks). Use of antibiotics in the past 6 weeks.
* Allergy to Fluorescein, Xylocaine or Propofol
* Known celiac disease
* Following a diet interfering with the study diet in opinion of the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Responder rates in targeted diet vs sham diet | After 4 weeks of dietary intervention
  Response defined by an improvement of minimum 50 points in the IBS-SSS.

SECONDARY OUTCOMES:
Baseline permeability measures between groups | At baseline
  Differences in baseline permeability measures between CLE positive and negative patients and healthy volunteers using Ussing chambers
Evolution of permeability measures between dietary interventions | Baseline and end of respective dietary intervention
  Differences in permeability measures between dietary interventions (i.e. verum, sham, wheat and soy) during the dietary interventions using urinary Lactulose/Mannitol/Sucralose ratio
Baseline mucosal immune cell composition between groups | Baseline
  Differences in baseline mucosal mast-cell and eosinophil counts between CLE positive and negative patients

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No